CLINICAL TRIAL: NCT05702346
Title: A Multi-level Telehealth Intervention to Enhance Physical Activity in Low-income Black and Hispanic Adults
Brief Title: Enhance Physical Activity in Low-income Black and Hispanic Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Simone V. Gill, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PA20183
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Physical Activity
Keywords: exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive the EPA intervention.
  Interventions: Behavioral: Enhance Physical Activity (EPA)
- Control (Active Comparator): This is the control group who will receive written information about health.
  Interventions: Behavioral: Enhance Physical Activity (EPA)

INTERVENTIONS:
Behavioral: Enhance Physical Activity (EPA) — EPA is eight weeks with four weekly, hour-long parts: virtual group exercises, virtual group discussions, individual PA participation, and individual phone check-ins.

SUMMARY:
The present study aims to test the efficacy of a multi-level telehealth intervention to Enhance Physical Activity (EPA) in 300 low-income Black and Hispanic/Latino adults. EPA is eight weeks with four weekly, hour-long parts: virtual group exercises, virtual group discussions, individual PA participation, and individual phone check-ins. A control group will receive health education. The specific aims are to: 1) test if physical activity increases significantly more among participants assigned to EPA vs. wait-list controls and 2) test if physical function improves significantly more among participants in EPA vs. controls. An exploratory third aim will test mechanisms of change associated with EPA.

DETAILED DESCRIPTION:
In the U.S., 77% of Black and 79% of Hispanic/Latino (HLs) adults do not meet physical activity (PA) guidelines to engage in moderate to vigorous PA for 150 minutes each week compared to 73% of White adults. Low PA leads to chronic conditions such as cardiovascular disease, type 2 diabetes, and obesity that result in disability and premature death. For Black and HL adults, low PA compounds predispositions to these conditions. Despite the urgent need to increase PA among Black and HL adults, solutions to increase PA are not tailored to this population. Poverty is more than double for Black (19.5%) and HLs (17%) compared to non-HL White adults (8.2%) and meeting PA standards increases with income. Lack of access to costly exercise facilities and living in unsafe neighborhoods contribute to low PA among Black and HL adults. As an alternative to traditional approaches, virtual guidance (i.e., telehealth) is a feasible and effective way to overcome the lack of access to facilities and PA participation in unsafe environments. The present study aims to test the efficacy of a multi-level telehealth intervention to Enhance Physical Activity (EPA) in 300 low-income Black and HLs. This full-scale, well-powered efficacy study builds on a Phase 1 pilot-controlled trial of EPA that showed high feasibility and acceptability in low-income Black and HLs. EPA is eight weeks with four weekly, hour-long parts: virtual group exercises, virtual group discussions, individual PA participation, and individual phone check-ins. Using a socio-ecological model of behavior change, EPA addresses PA and physical function at both intrapersonal (individual PA participation and individual phone check-ins) and interpersonal (virtual group exercises and virtual group discussions) levels. A control group will receive health education with the option to receive EPA later. All participants will attend four visits: pre-test, post-test 1 after EPA, post-test 2 (6 months after post-test 1), and post-test 3 (12 months after post-test 1). EPA is unique compared to other PA interventions as it combines standard PA intervention components with factors vital for increasing PA in Black and HLs while leveraging social connection: culturally relevant support, group discussions targeting discrimination, a telehealth format accessible to low-income people, and activities using everyday items or body weight to account for lack of equipment. The specific aims are to: 1) test if PA increases significantly more among participants assigned to EPA vs. wait-list controls and 2) test if physical function improves significantly more among participants in EPA vs. controls. An exploratory aim is to test mechanisms of change associated with EPA. Based on the sociocultural component of the National Institute on Minority Health and Health Disparities Research Framework, we hypothesize that social connection will mediate PA and physical function outcomes for those who receive the EPA intervention. This research can elucidate behavioral mechanisms responsible for low PA in low-income Black and HL adults and lead to scalable and sustainable multi-level interventions to support increased PA for Black and HL communities.

ELIGIBILITY:
Inclusion Criteria:

* being between 40-70 years old
* ability to speak and read English or Spanish
* ability to comply with study procedures and schedule
* having <150 minutes of weekly physical activity
* willingness to give informed consent

Exclusion Criteria:

* not independently ambulatory
* having other serious health problems that would make it difficult to participate for the duration of the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Physical activity | 12 months
  physical activity via the Physical Activity Scale for the Elderly
Objectively measured Physical activity | 12 months
  accelerometers
Physical function | 12 months
  physical function via the Short Physical Performance Battery

SECONDARY OUTCOMES:
Social determinants of health | 12 months
  surveys from the PhenX toolbox
Social connection | 12 months
  Social Connectedness questionnaire
Strength | 12 months
  strength with a hand-held dynamometer

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with any interested parties and will be disseminated via conferences.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All scientific data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: There are no anticipated factors or limitations that will affect the access, distribution or reuse of the de-identified scientific data generated by the study.